CLINICAL TRIAL: NCT07399847
Title: Effects of Time-of-day and Menstrual Cycle Phase (Low and High Progesterone) on Female's Cognitive and Strength Performance
Brief Title: Investigating the Effects of Time-of-day and Menstrual Cycle Phase (Low and High Progesterone) on Female's Cognitive and Strength Performance
Status: Not yet recruiting | Type: Observational
Sponsor: Lancaster University (Other)
Collaborators: Liverpool John Moores University (Other)
Responsible Party: Principal Investigator, Dr. Chris Gaffney, Senior Lecturer in Integrative Physiology, Lancaster University
Other Study IDs: FHM-2025-5797-RECR-2
Record Dates: First submitted 2026-01-13; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Circadian Rhythm; Menstrual Cycle Phase; Female Athletes; Executive Function (Cognition); Eumenorrhea; Strength

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Participants will have 90ml of bloods taken from their arm over the course of the study to measure levels of progesterone (P2), oestrogen (E2), inflammatory markers (Interleukin 6 (IL-6), Tumour necrosis factor alpha (TNF-alpha) and High-sensitivity C-reactive protein (hsCRP)) and for omics analysis.
  The blood will be centrifuged down and blood serum will be analysed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Female participants: Female (assigned at birth), aged 18-30 years. They must be tier 2 athletes which requires the participants to identify with a sport, train with a purpose to compete, regularly train ~3 times per week and compete at a local level. The participants must have a regular menstrual cycle - considered between 21-35-day cycles with at least 9 periods a year.
  Participants must not be currently/previously (in the last 3 months) using of any contraceptive method that alter the menstrual cycle or used the emergency contraceptive pill either 3 months prior to the study or during the study.

SUMMARY:
This study is designed to determine whether time-of-day and menstrual cycle phase influence athletic performance and is expected to contribute valuable insight into how both time-of-day, and hormonal factors can influence performance and expand existing research. This study aims to support more inclusive, effective and personalised approaches to training and competition schedules for female athletes.

The study will involve two testing days that require a participant to complete a compilation of tests at 07:00, 12:00 and 18:00 hours. The testing days will be arranged for when a participant is in phase 1 (lowest levels of progesterone in the menstrual cycle) and phase 4 (highest level of progesterone in the menstrual cycle). The tests will examine a participant's executive function and physical strength.

This study will aim to recruit thirty 18-30-year-old females from Lancaster University who identify with a sport that they train ~3 times a week for with a purpose to compete. The females recruited must have a regular menstrual cycle and no history of sleep disorders.

Aim: To investigate the effects of time-of-day and menstrual cycle phase (low and high progesterone levels) on executive function and strength in females.

Objectives:

1. To determine the effects of time-of-day on executive function and strength tests.
2. To determine the effects of menstrual cycle phase on executive function and strength tests.
3. To examine if there is an interaction between time-of-day and menstrual cycle phase on executive function and strength tests.

ELIGIBILITY:
Inclusion Criteria:

* Female (assigned at birth)
* Aged 18-30 years
* Tier 2 athlete which requires the participants to identify with a specific sport, train with a purpose to compete, regularly train ~3 times per week and compete at a local level (for example being a member of a BUCS sport and competing regularly with that sport)
* Regular menstrual cycle - considered between 21-35-day cycles with at least 9 periods a year.

Exclusion Criteria:

* The current/previous (in the last 3 months) use of any contraceptive method that alter the menstrual cycle
* The use of the emergency contraceptive pill either 3 months prior to the study or during the study
* Diagnosis of menstrual disorders including (but not exclusively) endometriosis and Polycystic Ovary Syndrome (PCOS)
* A formal diagnosis of sleep disorders such as insomnia
* Consume >400mg/day of caffeine
* A musculoskeletal injury in the past 3 months
* A formal diagnosis of neurological or psychiatric disorders such as Attention-Deficit/Hyperactivity Disorder (ADHD), Autism Spectrum Disorder (ASD), Dyslexia or schizophrenia
* Taking prescribed medication that may affect sleep for example stimulants such as Methylphenidate
* No regular night shift work
* No trans-meridian travel within 10 days of their expected participation dates (travel that will cause jetlag)
* Have given blood in the last 12 weeks - this is not strictly an exclusion; participants will just need to wait until after 12 weeks before taking part in the study

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will be selected from across Lancaster University (staff and students)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in muscle strength with time-of-day and menstrual cycle phase | 07:00, 12:00 and 18:00 hours in phase 1 and 4 (the points of low and high progesterone) of the menstrual cycle (each cycle is 21-35 days). Phase 1 is during menstruation and phase 4 is +7 days (±1) after the confirmation of the luteinising hormone peak.
  Repeated measures of strength at 07:00, 12:00 and 18:00 hours in phase 1 and 4 of the menstrual cycle. Handgrip strength requires participants to maximally squeeze the dynamometer for 3-seconds. 3 repeats will be carried out with the participants dominant hand, with 1-minutes of rest between each, recording the maximal values to determine both peak and mean values. Participants would also perform both countermovement and squat jumps, measuring flight time (seconds) and vertical jump height (centimetres). Each jump type will be repeated 3 times with a rest interval of 30-seconds between each jump repetition and a 2-minute rest interval between jump types. Maximal isometric Voluntary contraction of knee extensors and flexors would be measured over 4-seconds at 60° flexion. Between away and towards contractions, participants will have 30-seconds and between each set, they will have 3-minutes passive recovery.

SECONDARY OUTCOMES:
Change in cognitive performance with time-of-day and menstrual cycle phase | 07:00, 12:00 and 18:00 hours in phase 1 and 4 (the points of low and high progesterone) of the menstrual cycle (each cycle is 21-35 days). Phase 1 is during menstruation and phase 4 is +7 days (±1) after the confirmation of the luteinising hormone peak.
  Repeated measures of cognitive performance at 07:00, 12:00 and 18:00 hours across phase 1 and 4 of the menstrual cycle. It will be assessed with a modified Eriksen Flanker task. The task is a measure of inhibition and cognitive flexibility asking participants to respond to a visual stimulus depending on what is displayed on the screen and the instructions given. This modified flanker task uses arrows displayed on a screen and asking participants to focus on the central arrow that is flanked by arrows to its left and right, either congruent or incongruent to the central arrow. Section 1 of the task assesses simple reaction time whilst section 2 assesses inhibition and cognitive flexibility. Reaction time and number of correct answers for congruent and incongruent sequences will be determined and analysed as an indicator of cognitive flexibility and inhibition (two measures of executive function).
Change in menstrual cycle symptoms with time-of-day and menstrual cycle phase | 07:00, 12:00 and 18:00 hours in phase 1 and 4 (the points of low and high progesterone) of the menstrual cycle (each cycle is 21-35 days). Phase 1 is during menstruation and phase 4 is +7 days (±1) after the confirmation of the luteinising hormone peak.
  During testing visits, questions will be asked regarding participants current menstrual symptoms to determine what affects their current phase of the menstrual cycle could be having on them. The questionnaire during testing will be repeated at 07:00, 12:00 and 18:00 hours across phase 1 and phase 4 of the menstrual cycle.
Ovulation phase confirmation | Prior to testing visit and the following menstrual cycle. The day to begin ovulation testing varies depending on menstrual cycle length (21-35 days) but typically will begin around day 10 of each cycle, with day 1 being the first day of bleeding.
  Participants will be asked to use ovulation strips three days before they are expected to ovulate and confirm with the researcher when they have had the positive test. They will carry out ovulation testing for two consecutive cycles of their menstrual cycle and report these both to the researcher. This study requires two testing visits to the lab, one when progesterone levels are at their lowest (during your period days 1-5) and one when progesterone levels are at their highest (just after ovulation typically around day 19-21). Participants will be asked to track their menstrual cycle on an app so that the researcher can arrange testing day visits.
Change in participant weight with time-of-day and menstrual cycle phase | 07:00, 12:00 and 18:00 hours in phase 1 and 4 (the points of low and high progesterone) of the menstrual cycle (each cycle is 21-35 days). Phase 1 is during menstruation and phase 4 is +7 days (±1) after the confirmation of the luteinising hormone peak.
  Participants weight (kilograms) will be taken at each visit to provide information about weight fluctuation across the menstrual cycle phases and time-of-day.
Change in hormone levels with time-of-day and menstrual cycle phase | 07:00, 12:00 and 18:00 hours in phase 1 and 4 (the points of low and high progesterone) of the menstrual cycle (each cycle is 21-35 days). Phase 1 is during menstruation and phase 4 is +7 days (±1) after the confirmation of the luteinising hormone peak.
  Participant will have their blood drawn at both visits (phase 1 and 4) and at all three times of the day (07:00, 12:00 and 18:00 hours). Over the course of the study, 90milliletres (ml) (~15 teaspoons) of blood will be collected - 15ml of blood at each visit (3 tubes of blood each 5ml in volume). The blood samples collected in vacutainers would be stored at -80°c before carrying out various assays on participant's blood serum (separated and collected following centrifugation), according to manufacturer's guidelines, to measure progesterone (P) and oestradiol (E2). Blood analysis of progesterone and oestrogen would be carried out in duplicate using commercially available serum and plasma enzyme linked immunosorbent assays (ELISA). The blood analysis would act to confirm correct phase identification during testing, with the exclusion of participants occurring after testing due to E2 or P levels not matching those defined for Phase 1 and 4.
Change in core body temperature with time-of-day and menstrual cycle phase | 07:00, 12:00 and 18:00 hours in phase 1 and 4 (the points of low and high progesterone) of the menstrual cycle (each cycle is 21-35 days). Phase 1 is during menstruation and phase 4 is +7 days (±1) after the confirmation of the luteinising hormone peak.
  Repeated measures of core body temperature will be measured at 07:00, 12:00 and 18:00 hours in phase 1 and 4 of the menstrual cycle, using a thermometer placed in the ear, two measures will be taken 2-minutes apart, if the difference between the values is >0.2°c then a third measure would be taken. The average temperature would be calculated as the mean of the closest pair of measurements. Core body temperature is a marker of circadian rhythm.
Change in blood pressure with time-of-day and menstrual cycle phase | 07:00, 12:00 and 18:00 hours in phase 1 and 4 (the points of low and high progesterone) of the menstrual cycle (each cycle is 21-35 days). Phase 1 is during menstruation and phase 4 is +7 days (±1) after the confirmation of the luteinising hormone peak.
  Repeated measures of blood pressure will be measured at 07:00, 12:00 and 18:00 hours in phase 1 and 4 of the menstrual cycle, using an automatic blood pressure monitor as a cross-validation method of core body temperature to determine circadian rhythm phase of each participant.
Change in heart rate variability with time-of-day and menstrual cycle phase | 07:00, 12:00 and 18:00 hours in phase 1 and 4 (the points of low and high progesterone) of the menstrual cycle (each cycle is 21-35 days). Phase 1 is during menstruation and phase 4 is +7 days (±1) after the confirmation of the luteinising hormone peak.
  Repeated measures of hear rate variability will be measured at 07:00, 12:00 and 18:00 hours in phase 1 and 4 of the menstrual cycle. HRV is measured in both frequency and time domains, root mean square of successive differences (RMSSD), and high- and low-frequency (HF and LF) respectively. These measures indicate the balance between parasympathetic and sympathetic activity of the autonomic nervous system and have been shown to vary with time-of-day, and will be used as a cross-validation to determine a participants circadian rhythm phase.
Change in brain activity with time-of-day and menstrual cycle phase | 07:00, 12:00 and 18:00 hours in phase 1 and 4 (the points of low and high progesterone) of the menstrual cycle (each cycle is 21-35 days). Phase 1 is during menstruation and phase 4 is +7 days (±1) after the confirmation of the luteinising hormone peak.
  Repeated measures of brain activity using an 8-lead Electroencephalography (EEG) system to analyse neural activity at resting-state will be carried out at 07:00, 12:00 and 18:00 hours in phase 1 and 4 of the menstrual cycle. The sliver-silver chloride (Ag|AgCl) electrodes are prepositioned (Cz, F3, F4, Pz, P7, P8, O1 and O2) according to the international 10-20 montage system in a head cap that is placed on the participants head prior to recording. Participants will relax for 2-minutes with ear plugs and eyes closed to reduce the level of external stimuli. The first EEG recording is for 5-minutes with eyes closed, the second recording is eyes open for 5-minutes focusing on a black cross on a white background and the third recording will take place during the Flanker task. EEG power in alpha and theta bands will be analysed. Participants will not be told how long each recording is for as they will be asked to answer questions regarding this time as another measure (temporality).
Changes in temporality with time-of-day and menstrual cycle phase | 07:00, 12:00 and 18:00 hours in phase 1 and 4 (the points of low and high progesterone) of the menstrual cycle (each cycle is 21-35 days). Phase 1 is during menstruation and phase 4 is +7 days (±1) after the confirmation of the luteinising hormone peak.
  Participants will be asked several temporal questions which focus on their perception of time, the questions will ask about the amount of time the participants spent with their eyes closed/open and if these times vary between different testing times (07:00 and 18:00 hours) and different phases (phase 1 compared to phase 4).
Changes in inflammatory markers with time-of-day and menstrual cycle phase | 07:00, 12:00 and 18:00 hours in phase 1 and 4 (the points of low and high progesterone) of the menstrual cycle (each cycle is 21-35 days). Phase 1 is during menstruation and phase 4 is +7 days (±1) after the confirmation of the luteinising hormone peak.
  Participant will have their blood drawn at both visits (phase 1 and 4) and at all three times of the day (07:00, 12:00 and 18:00 hours) (repeated measures). Over the course of the study, 90ml (~15 teaspoons) of blood will be collected - 15ml of blood at each visit (3 tubes of blood each 5ml in volume). Blood samples collected in vacutainers would be stored at -80°c before being centrifuged to collect blood serum for analysis using various assays, according to manufacturer's guidelines, to measure Interleukin (IL-6), Tumour necrosis factor (TNFα) and high sensitivity C reactive protein (hsCRP) levels. The blood analysis of common inflammatory markers (IL-6, TNF-α and CRP) on female tier 2 athletes will provide a greater understanding of biochemical interactions when considering the possible strength and cognitive performance fluctuations possibly observed with time-of-day and menstrual cycle.
Change in glucose and lactate blood levels in the morning with menstrual cycle phase | 07:00 hours in phase 1 and 4 of the menstrual cycle (each cycle is 21-35 days). Phase 1 is during menstruation and phase 4 is +7 days (±1) after the confirmation of the luteinising hormone peak.
  This measure will only be performed at the morning visit to consider blood glucose and lactate levels after the overnight fast. A small volume of blood will be taken from the vacutainers of blood collected and placed in a capillary tube to carry out glucose and lactate analysis of the participants in the morning in phase 1 and 4 of the menstrual cycle due to the possible effects of differing blood glucose levels on cognition.
Monitoring of participant diet intake | On the days of both testing visits, phase 1 and 4 of the menstrual cycle (each cycle lasting 21-35 days). Phase 1 is during menstruation and phase 4 is +7 days (±1) after the confirmation of the luteinising hormone peak.
  Participants will be provided with a food diary to track what they ate on the day of their first testing visit to record what time they ate and what they consumed so that they can ensure they consume identical meals at identical mealtimes when it comes to their second visit, acting as a control measure.
Changes in sleep quality with menstrual cycle phase | 07:00 hours across phase 1 and 4 of the menstrual cycle (each cycle 21-35 days). Phase 1 is during menstruation and phase 4 is +7 days (±1) after the confirmation of the luteinising hormone peak.
  During testing visits, questions will be asked regarding the participants quality of sleep from the night before each testing visit (phase 1 and 4 of the menstrual cycle) to determine what affects their quality of sleep could be having on them. The questionnaire during testing will be carried out at 07:00 hours across phase 1 and phase 4 of the menstrual cycle.
Changes in mood states with time-of-day and menstrual cycle phase. | 07:00, 12:00 and 18:00 hours across phase 1 and 4 of the menstrual cycle (cycle of 21-35 days). Phase 1 is during menstruation and phase 4 is +7 days (±1) after the confirmation of the luteinising hormone peak.
  During testing visits, questions will be asked regarding participants current mood state using a profile of mood states questionnaire (POMS) to determine what affects this could be having on them. The questionnaire during testing will be repeated at 07:00, 12:00 and 18:00 hours across phase 1 and phase 4 of the menstrual cycle.
Changes in caffeine withdrawal symptoms with time-of-day and menstrual cycle phase. | 07:00, 12:00 and 18:00 hours across phase 1 and 4 of the menstrual cycle (each cycle is 21-35 days). Phase 1 is during menstruation and phase 4 is +7 days (±1) after the confirmation of the luteinising hormone peak.
  During testing visits, questions will be asked regarding participants current experiences of caffeine withdrawal to determine what effects this could be having on them. The questionnaire during testing will be repeated at 07:00, 12:00 and 18:00 hours across phase 1 and phase 4 of the menstrual cycle.
Screening of general health to ensure eligibility | The familiarisation visit will take place 1-2 weeks before the testing visit. Whether a participant is tested in phase 1 or 4 (this is randomised) will dictate when the familiarisation visit will occur.
  With the use of questionnaires, participants will be asked questions prior to the testing visits regarding their general health (American college of sports medicine participant health screening (ACSM)). This is to confirm their eligibility with regards to health for the study.
Screening for menstrual cycle irregularities to confirm eligibility. | The familiarisation visit will take place 1-2 weeks before the testing visit. Whether a participant is tested in phase 1 or 4 (this is randomised) will dictate when the familiarisation visit will occur.
  With the use of questionnaires, participants will be asked questions prior to the testing visits regarding their menstrual cycle health (menstrual distress questionnaire (MEDI-Q) and additional questions regarding cycle regularity). This is to confirm their eligibility with regards to their menstrual cycle for the study.
Determination of participant chronotype. | The familiarisation visit will take place 1-2 weeks before the testing visit. Whether a participant is tested in phase 1 or 4 (this is randomised) will dictate when the familiarisation visit will occur.
  With the use of questionnaires, participants will be asked questions prior to the testing visits regarding their sleep-wake habits (the composite morningness questionnaire). This is to determine participants chronotype (morning or evening person) prior to the start of the study.
Screening of participants caffeine consumption to ensure eligibility | The familiarisation visit will take place 1-2 weeks before the testing visit. Whether a participant is tested in phase 1 or 4 (this is randomised) will dictate when the familiarisation visit will occur.
  With the use of questionnaires, participants will be asked questions prior to the testing visits regarding their daily caffeine consumption. This is to confirm their eligibility with regards to caffeine consumption for the study.

DOCUMENTS (2):
  • Study Protocol (2026-01-05): https://cdn.clinicaltrials.gov/large-docs/47/NCT07399847/Prot_000.pdf
  • Informed Consent Form (2026-01-05): https://cdn.clinicaltrials.gov/large-docs/47/NCT07399847/ICF_001.pdf